CLINICAL TRIAL: NCT05246371
Title: Propofol/Dexmedetomidine Versus Desflurane Effects on Post Hepatectomy Hepatocellular Injury
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ain Shams anesthesia Dep
Record Dates: First submitted 2022-01-21; First posted 2022-02-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Hepatectomy
MeSH Terms: interventions — Propofol; Dexmedetomidine; Desflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- propofol and dexmedetomidine (Experimental): Patients will receive maintenance of general anesthesia by TIVA using combination of propofol and dexmedetomidine
  Interventions: Drug: Propofol, dexmedetomidine
- desflurane (Experimental): Patients will receive maintenance of general anesthesia by desflurane.
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Propofol, dexmedetomidine — Patients will receive maintenance of general anesthesia by TIVA using combination of propofol and dexmedetomidine.
  Other Names: TIVA
  Arms: propofol and dexmedetomidine
Drug: Desflurane — Patients will receive maintenance of general anesthesia by desflurane.
  Other Names: inhalational anesthesia
  Arms: desflurane

SUMMARY:
This study will compare the effects of propofol/dexmedetomidine versus desflurane for maintenance of general anesthesia on hepatocellular injury in patients undergoing partial hepatectomy.

DETAILED DESCRIPTION:
Postoperative impairment of liver function is common after hepatectomy. It may be caused by surgical trauma, loss of hepatic mass, stress response, hepatic oxygen deprivation, infection and drug toxicity.

Anesthetic agents used in general anesthesia for liver surgery have a big effect on hepatic blood flow, oxygen delivery and liver function This study will compare the effects of propofol/dexmedetomidine versus desflurane for maintenance of general anesthesia on hepatocellular injury in patients undergoing partial hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of Anesthesiologists physical status (ASA) I to II.
2. Patients Child Pugh classification A to B.
3. Both sexes.
4. Aged between 18 years and 70 years
5. Scheduled for more than 1 segment hepatectomy.

Exclusion Criteria:

1. Patients with Child Pugh classification C.
2. Patients younger than18 years old or older than 70 years old
3. Patients performed additional ablation therapies (cryosurgery or radiofrequency ablation).
4. Prior liver resection for donation.
5. Scheduled resection not requiring inflow occlusion (Pringle's maneuver).
6. Hypersensitivity to any of the used drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
aspartate aminotransferase (AST) | 1 week
  aspartate aminotransferase (AST)
alanine aminotransferase (ALT) | 1 week
  alanine aminotransferase (ALT)
bilirubin | 1 week
  bilirubin
albumin | 1 week
  albumin
prothrombin time | 1 week
  prothrombin time
INR | 1 week
  INR

CONTACTS AND LOCATIONS:
Overall Officials: Hany Alzahaby, Professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
open source
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: open source